CLINICAL TRIAL: NCT03000023
Title: A Qualitative and Quantitative Evaluation of Patients' Anticipated and Perceived Treatment Benefits Following HCV Viral Eradication
Brief Title: Anticipated and Perceived Benefits Following Hepatitis C Treatment
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: 15-2081
Record Dates: First submitted 2016-12-06; First posted 2016-12-21 (Estimated); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Hepatitis C; Hepatitis C, Chronic
Keywords: Hepatitis C; Patient-Reported Outcomes; DAA Treatment; Qualitative; Mixed methods
MeSH Terms: conditions — Hepatitis C; Hepatitis C, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The study is both qualitative and quantitative, gathering patient's perceptions of HCV treatment benefits before and after HCV treatment by administering surveys and conducting in-depth qualitative patient interviews. The study seeks to understand all anticipated and actual benefits patients perceive before and after viral eradication.

DETAILED DESCRIPTION:
This study employs a mixed methods (qualitative and quantitative) pre-post study design utilizing in-depth qualitative interviews and patient reported outcome surveys. Pre-treatment surveys and interviews will be conducted before HCV therapy commences to understand all potential psychological, social, physical and medical consequences perceived to be related to HCV and the patients' anticipation (hope for) of improvements in these factors after viral eradication. Post-treatment surveys and interviews will occur 4 to 8 months after treatment ends to examine long-term treatment benefits, i.e., changes in HCV-related factors, such as symptoms, functioning, and health status.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 or older
* English-speaking
* Any genotype
* Any treatment duration (e.g. 8, 12, or 24 weeks)
* Has been written a prescription for a sofosbuvir (SOF)-containing regimen.

Exclusion Criteria:

* Currently listed for liver transplant; post-liver transplant

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Hepatitis C
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-10; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Analyze changes in patient perceptions through qualitative interviews before and after HCV treatment. | 1 Year
  To conduct a pre-post qualitative analysis that will evaluate changes in a broad range of patients' perceptions of psychological, social, and physical effects associated with HCV and viral cure collected through qualitative interviews.
Evaluate pre-post survey change in patient reported HCV symptoms and other factors. | 1 Year
  To conduct a pre-post survey evaluation of change in patient-reported HCV symptoms, functioning, and health perceptions associated with HCV and viral cure.

CONTACTS AND LOCATIONS:
Overall Officials: Donna Evon, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No